CLINICAL TRIAL: NCT04571021
Title: Implementation of the Individual Danish Emergency Process Triage (I-DEPT)
Brief Title: Implementation of the Individual Danish Emergency Process Triage
Acronym: I-DEPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Collaborators: Amager Hospital (Other); University Hospital Bispebjerg and Frederiksberg (Other); Nykøbing Falster Hospital, Department of Emergency Medicine (Unknown); Slagelse Hospital, Department of Emergency Medicine (Unknown); Køge Hospital, Department of Emergency Medicine (Unknown); Nordsjaellands Hospital (Other); Holbæk Hospital, Department of Emergency Medicine (Unknown)
Responsible Party: Principal Investigator, Kasper Iversen, Professor, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 568
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Acute Disease; Emergencies; Clinical Syndrome
Keywords: triage; risk stratification; emergency department
MeSH Terms: conditions — Acute Disease; Emergencies

STUDY DESIGN:
Intervention Model Description: Stepped-Wedge cluster randomized design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-DEPT (Experimental): Novel triage. The triage nurse can adjust the triage category one level of urgency down or one or two levels up.
  Interventions: Other: I-DEPT
- DEPT (Active Comparator): Existing triage algorithm
  Interventions: Other: DEPT

INTERVENTIONS:
Other: I-DEPT — Implementation of the novel triage algorithm
  Arms: I-DEPT
Other: DEPT — Existing triage algorithm
  Arms: DEPT

SUMMARY:
The purpose of the study is to implement and evaluate a novel triage algorithm for risk stratification of acutely admitted patients in the Emergency Department.

DETAILED DESCRIPTION:
Triage algorithms are used worldwide to risk assess and prioritize patients in the Emergency Departments. The aim is to identify patient at risk of deterioration or death and/or with a imminent need of treatment. The triage algorithms are also developed to identify patients at low risk, who safely can be assigned to the waiting room.

Currently, several different triage algorithms are used, and they are mostly based on consensus and exper- opinion. Therefore evidence concerning triage is limited.

The investigators has developed a novel evidence-based triage algorithm with integrated individual clinical assesment. The vitals measured at admission assigns the patient to a triage category, and based upon the clinical appearance of the patients, the triage nurse can adjust the assigned triage category to better reflect the patient. The triage algorithm used in Denmark is "DEPT", this algorithm is based purely on vitals and cause of admission and can not be adjusted.

I-DEPT is designed as a cluster randomized stepped-wedge non-inferiority study. The Aim is to implement and compare I-DEPT to the existing triage algorithm. All Emergency Departments in the Capitol Region and the Region og Zealand in Denmark will implement I-DEPT one department at a time (8 centers). The first will start the implementation on october 1, 2020 and after two months the next center will implement I-DEPT. Every two months a new center will start. During 16 months all centers will have implemented I-DEPT the sequence of centers was determined by randomization. The first 30 days of implementation will be censored and not included in the final analyses. The study will conclude with a period of 30 days follow-up. Patients will only be included once.

ELIGIBILITY:
Inclusion Criteria:

* Admission to a participating Emergency Department in the study period
* Full triage assesment in the index admission

Exclusion Criteria:

* Age below 17 years
* Death at arrival or before triage assesment

Ages: 17 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250000 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
30-day mortality | 30 days
  All cause mortality within 30 days following triage in the index admission by non-inferiority

SECONDARY OUTCOMES:
2-day mortality | 2 days
  All cause mortality within 2 days following triage in the index admission
Distribution of triage categories | 1 day
  There are four categories in both triage algorithms used in this study: (green (least urgent), yellow, orange, and red (most urgent))
Patients in the orange triage category | 1 day
  Number of patients assigned to the orange category
Doctor assessment | 1 day
  Time from triage to arrival of a doctor
Days in hospital | 30 days
  The number of days admitted to a hospital within 30 days
Time in the Emergency Department | 30 days
  Time spent in the Emergency department from triage to either admission, transfer or discharge
Patients left without being seen | 30 days
  Number of patients leaving the Emergency Department without being assessed by a doctor

CONTACTS AND LOCATIONS:
Overall Officials: Kasper K Iversen, Professor, Principal Investigator — Herlev and Gentofte Hospital
Locations (8):
- Denmark (8):
  - Herlev and Gentofte hospital, Herlev, Capital Region
  - Bispebjerg and Frederiksberg hospital, Copenhagen
  - Nordsjællands Hospital, Hillerød
  - Holbæk hospital, Holbæk
  - Hvidovre, Amager and Glostrup Hospital, Hvidovre
  - Sjælland University hospital, Køge
  - Nykøbing Falster Hospital, Nykøbing Falster
  - Slagelse Hospital, Slagelse

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/21/NCT04571021/SAP_000.pdf